CLINICAL TRIAL: NCT00505167
Title: Memantine Versus Donepezil in Mild to Moderate Alzheimer's Disease. A Randomized Trial With Magnetic Resonance Spectroscopy.
Brief Title: Memantine Versus Donepezil in Early Stages of Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Clinica Quiron de Zaragoza (Unknown); Universidad de Zaragoza (Other); Hospital de Barbastro (Unknown); Hospital Royo Villanova (Unknown)
Responsible Party: Dr Pedro J Modrego, Department of Neurology. hospital Miguel Servet. Zaragoza. Spain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0910-0459
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Dementia, Alzheimer Type
Keywords: Alzheimer's disease; Memantine; Donepezil; Magnetic resonance Spectroscopy; randomized trial
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine; Donepezil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients randomized to receive memantine
  Interventions: Drug: Memantine
- 2 (Active Comparator): Patients randomized to receive donepezil
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Memantine — Patients randomized to receive either memantine or donepezil
  Other Names: Ebixa (Memantine)
  Arms: 1
Drug: Donepezil — Patients randomized to receive either memantine or donepezil
  Other Names: Aricept (Donepezil)
  Arms: 2

SUMMARY:
It is well known that in the brain of the patients with Alzheimer's disease there is a glutamatergic hyperstimulation leading to neuronal death. Memantine is a low affinity antagonist of NMDA glutamate receptors. The use of this drug in the early phases of the disease could provide neuroprotective effects and delay of progression. The effects of memantine should be compared to those of donepezil, which is the most prescribed anticholinesterase drug.

DETAILED DESCRIPTION:
On the basis of the excess of glutamatergic stimulation, our objective is to demonstrate whether memantine could have a neuroprotective effect in Alzheimer's disease when administered in the early stages and in comparison to donepezil. The patients would be randomized to receive one of these drugs. At baseline we would evaluate the patients from a clinical standpoint with the ADAS-cog, the neuropsychiatric Inventory and a scale of daily living activities.We also would carry out Magnetic Resonance Spectroscopy in several areas of the brain (medial temporal lobe, prefrontal region, cingulate gyrus and occipital lobe) so as to measure the concentration of N-acetyl-aspartate which is a marker of neuronal density.Then we treat the patients with either memantine or denepezil and after 6 months we would repeat the same procedures as we did at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria of probable Alzheimer's disease in the stages mild-to-moderate with a Mini-Mental score higher than 15 points.

Exclusion Criteria:

* Previous treatment with anticholinesterase drugs or memantine.
* Advanced stages of the disease
* Lack of a reliable caregiver.
* Dementias other than Alzheimer's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in the Levels of the metabolite N-acetyl-aspartate in several areas of the brain. | 6 months

SECONDARY OUTCOMES:
Changes in the clinical scales observed after treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Modrego, MD, Principal Investigator — Department of Neurology. Hospital Miguel Servet. Zaragoza. Spain
Locations (3):
- Spain (3):
  - Hospital de Barbastro, Barbastro, Huesca
  - Cenro de especialidades San José. Hospital Miguel Servet, Zaragoza
  - Hospital Royo Villanova, Zaragoza

REFERENCES:
- [Derived] Modrego PJ, Fayed N, Errea JM, Rios C, Pina MA, Sarasa M. Memantine versus donepezil in mild to moderate Alzheimer's disease: a randomized trial with magnetic resonance spectroscopy. Eur J Neurol. 2010 Mar;17(3):405-12. doi: 10.1111/j.1468-1331.2009.02816.x. Epub 2009 Oct 28. PMID 19874395